CLINICAL TRIAL: NCT07374861
Title: Multicenter Study on the Evaluation of Adherence, Persistence and Efficacy of Treatment With Bempedoic Acid in Italy
Acronym: BEMPENET
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Pasquale Perrone Filardi, Professor, Federico II University
Other Study IDs: Prot. 28/2025
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with hyperlipidaemia under Bempedoic acid treatment
  Interventions: Drug: Bempedoic acid

INTERVENTIONS:
Drug: Bempedoic acid — film-coated tablets

SUMMARY:
Evaluation of adherence, persistence, and efficacy of treatment with Bempedoic acid in a real-life Italian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients under Bempedoic acid treatment

Exclusion Criteria:

* Age < 18 years o > 80 years
* Patients who refuse to participate and to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients from Italy who have received Bempedoic acid as part of routine clinical management of their hyperlipidaemia, based on national reimbursement criteria at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Description of adherence to treatment with Bempedoic acid in a real-life Italian population | 6-12-24-36 months
  Adherence will be assessed in terms of Medical Possession Ratio (MPR), which is defined as the ratio between the treatment units dispensed during the treatment period and the duration of the treatment period itself.
Description of efficacy of treatment with Bempedoic acid in a real-life Italian population | 6-12-24-36 months
  Efficacy of treatment will be evaluated as a change in the LDL (deltaLDL) value from the start of treatment (percentage and absolute value).
Description of persistence to treatment with Bempedoic acid in a real-life Italian population | 6-12-24-36 months
  Persistence will be assessed in terms of therapeutic continuity from the start of treatment to enrollment.

SECONDARY OUTCOMES:
Description of safety of treatment with Bempedoic acid in a real-life Italian population | 6-12-24-36 months
  Safety will be evaluated in terms of adverse reactions or intolerance to the drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University of Naples, Department of Advanced Biomedical Sciences, Napoli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No